CLINICAL TRIAL: NCT06131476
Title: Clinical Investigation of Visual Acuity in Contact Lens Wearers After Instillation of a Lipid- Based Lubricating Eye Drop
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6371
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Test/Control sequence, to receive the TEST lubricating eye drops, with a washout period of 90 minutes between instillations. After the wash-out period, the CONTROL lubricating eye drops will be instilled.
  Interventions: Drug: Blink® Tears eye drops; Drug: Investigational lipid eye drops
- Control/Test (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomized into the Test/Control sequence, to receive the CONTROL lubricating eye drops, with a washout period of 90 minutes between instillations. After the wash-out period, the TEST lubricating eye drops will be instilled.
  Interventions: Drug: Blink® Tears eye drops; Drug: Investigational lipid eye drops

INTERVENTIONS:
Drug: Blink® Tears eye drops — Control Drops
Drug: Investigational lipid eye drops — Test Drops

SUMMARY:
This is a single visit, randomized, double masked, bilateral, non-dispensing, 2×2 crossover study to assess visual acuity.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Between 18 and 69 (inclusive) years of age at the time of screening.
4. Subjects must be habitual spherical soft contact lens wearers.
5. Subjects must achieve visual acuity of 20/30 or better in each eye with their habitual contact lenses.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

The subject must not:

1. Currently pregnant or breast-feeding.
2. Diabetes.
3. Any ocular or systemic allergies or disease which may interfere with the clinical trial (at the discretion of the investigator).
4. Any systemic disease, autoimmune disease, or use of medication which may interfere with the clinical trial (at the discretion of the investigator).
5. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self-report.
6. History of any ocular or corneal surgery (e.g. RK, PRK, LASIK)
7. Participation in any pharmaceutical or medical device related clinical trial within 14 days prior to study enrollment.
8. History of binocular vision abnormality or strabismus.
9. Habitual wearers of rigid gas permeable lens within the past 3 months5. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g., SynergEyes, SoftPerm) within the past 6 months.
10. Current habitual use of Prescription Medication to treat dry eye or ocular discomfort, ocular steroids, or any medication (RX or OTC) that would interfere with the clinical study (at the discretion of the investigator)
11. Employees of investigational clinic (investigator, coordinator, and technician etc) or family members of an employee of the clinical site by self-report.
12. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, cornea vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale.
13. Any active ocular abnormalities/conditions that may interfere with the clinical trial (this includes, but not limited to, chalazia, recurrent styles, pterygium, infection, etc.).
14. Any corneal distortion due to previous rigid gas permeable lens wear, surgery or pathology.\ In addition to the above criteria, patients with any allergy or sensitivity to ingredients that this product may contain should not participate in the study (Castor Oil, Polyoxyl 40 Hydrogenated Castor Oil, Sodium Chlorite, Boric Acid, Sodium Borate Decahydrate, Sodium Chloride, Potassium Chloride, Calcium Chloride Dihydrate, Magnesium Chloride Hexahydrate, Polyethylene Glycol 400, Sodium Hyaluronate, Purified Water).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (2):
- United States (2):
  - Vue Optical Boutique, Jacksonville, Florida
  - St. Johns Eye Associates, P.A., Saint Augustine, Florida

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 32 subjects were enrolled from two clinical sites in this study. Of those enrolled, a total of 31 (96.9%) subjects were randomly assigned among 2 unique eye drop sequences, study eye drops administered in both eyes for all subjects and were included in Safety Population; while, one (3.1%) subject was a screen failure and/or not assigned. Of the total assigned subjects, all 31 (96.9%) subjects completed the study.
Groups:
- Investigational Lipid Drop\Blink Tears: Subjects randomized to this sequence received Investigational Lipid Drop during the first period and then received Blink Tears during the second period
- Blink Tears\Investigational Lipid Drop: Subjects randomized to this sequence received Blink Tears during the first period and then received Investigational Lipid Drop during the second period
Period: Period 1
Arm/Group | Investigational Lipid Drop\Blink Tears | Blink Tears\Investigational Lipid Drop
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Investigational Lipid Drop\Blink Tears | Blink Tears\Investigational Lipid Drop
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who instilled at least one eye drop
Groups:
- Total: All subjects who instilled at least one eye drop.
Arm/Group | Total
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.9 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 3
  Black or African American | 1
  White | 26
  Other | 1
Region of Enrollment [Number; unit: Participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity (logMAR) at 3 Minutes Post Instillation
Description: High contrast bright illumination monocular logMAR (Logarithm of the Minimum Angle of Resolution) visual acuity was assessed at distance (4 meters) using ETDRS Charts, near (40 cm) and intermediate (64 cm) using reduced Guillon-Poling charts. A value of 0.0 logMAR indicated a Snellen vision of 20/20. Lower logMAR visual acuity values indicate better vision. The average logMAR visual acuity for each treatment was reported.
Time Frame: 3 minutes post instillation
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Groups:
- Investigational Lipid Drop: Subjects who instilled the Investigational Lipid Drop in the first or second period of the study.
- Blink Tears: Subjects who instilled the Blink Tears in the first or second period of the study.
Arm/Group | Investigational Lipid Drop | Blink Tears
Number analyzed (Participants) | 31 | 31
Number analyzed (Eyes) | 62 | 62
LogMAR | 0.09 (0.082) | 0.08 (0.088)

2. Primary Outcome: Visual Acuity (logMAR) at 10 Minutes Post Instillation
Description: as for outcome 1
Time Frame: 10 minutes post instillation
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: Eyes
Arm/Group | Investigational Lipid Drop | Blink Tears
Number analyzed (Participants) | 31 | 31
Number analyzed (Eyes) | 62 | 62
LogMAR | 0.09 (0.095) | 0.09 (0.087)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject is approximately 3 hours within 1 day.
Arm/Group | Investigational Lipid Drop | Blink Tears
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT06131476/Prot_SAP_000.pdf